CLINICAL TRIAL: NCT02329717
Title: A Phase II, Single-arm, Open-label, Bayesian Adaptive Efficacy and Safety Study of PBI-05204 in Patients With Stage IV Metastatic Pancreatic Adenocarcinoma
Brief Title: Efficacy and Safety Study of PBI-05204 in Patients With Stage IV Metastatic Pancreatic Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phoenix Biotechnology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-4350
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PBI 05204 (Experimental): PBI 05204 capsules dosed at 0.2255 mg/kg/day, continuous dosing
  Interventions: Drug: PBI 05204

INTERVENTIONS:
Drug: PBI 05204 — PBI 05204 daily dosing

SUMMARY:
This study evaluates the efficacy and safety of PBI-05204, an extract of the leaves of Nerium oleander, in patients with Stage IV metastatic pancreatic cancer. All patients will receive PBI-05204.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged ≥18 years.
2. Patient with histologically-confirmed Stage IV malignant metastatic adenocarcinoma of the pancreas; (a) who has relapsed from or is refractory to standard therapy and for whom no therapy exists that would be curative or might provide significant benefit or (b) who are intolerant to or refuse standard chemotherapy and, therefore, for whom experimental therapy is a reasonable option.
3. Patient has measurable disease, as determined by the Investigator using RECIST, version 1.1, as determined within 28 days before baseline (C1D1).
4. Patient has an ECOG performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), as assessed on C1D1, before the first dose of PBI 05204.
5. Patient has a predicted life-expectancy of ≥3 months.
6. Patient has adequate bone marrow function defined as:

   * Absolute neutrophil count (ANC) (neutrophil and bands) ≥1.5 x 10 ^9/L
   * Platelet count ≥100 x10^9/L
   * Hemoglobin ≥9.0 g/dL
7. Patient has adequate hepatic function defined as:

   * Total bilirubin within normal limits (WNL) for the institution, unless the bilirubin abnormality is considered due to Gilbert's syndrome.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.0 x the institutional upper limit of normal (ULN), or, in patients with known liver metastases, ≤5.0 x the institutional ULN.
   * Serum albumin ≥3.0 g/dL.
8. Patient has adequate renal function defined as:

   Serum creatinine ≤1.5 the institutional ULN
9. Patient has serum potassium and magnesium levels WNL for the institution and total serum calcium or ionized calcium levels ≥ the lower limit of normal (LLN). Patients with low potassium, calcium, and/or magnesium levels may receive supplementation to meet the protocol entry criteria. (Calcium supplementation is prohibited after starting PBI-05204; see Appendix 2.)
10. Patient provides signed and dated informed consent prior to initiation of any study procedures.
11. Patient and his/her partner agree to use adequate contraception after providing written informed consent through 3 months after the last dose of PBI 05204, as follows:

    * For women: Negative pregnancy test during screening (Day 3 to Day 1) before C1D1 and compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or postmenopausal (defined as amenorrhea for ≥12 consecutive months; or receiving hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level >35 mIU/mL).
    * For men: Compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile. Men whose sexual partners are of child-bearing potential must agree to use a medically-approved contraceptive regimen during the study and for 3 months after the treatment period.
12. Patient is capable of swallowing study drug capsules whole.
13. Patient is willing and able to participate in the study and comply with all study requirements.

Exclusion Criteria:

1. Patient has uncontrolled or significant cardiovascular disease, including:

   * Myocardial infarction within 6 months before C1D1.
   * Uncontrolled angina within 3 months before C1D1.
   * Congestive heart failure, defined as New York Heart Association (NYHA) Class II, within 3 months before C1D1 (see Appendix 1).
   * Diagnosed or suspected congenital long QT syndrome.
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White [WPW] syndrome, or torsade de pointes), or prolonged QTc interval on pre-entry ECG (>450 msec). If the automated reading is prolonged (i.e., >450 msec), the ECG should be manually over-read.
   * Any history of second- or third-degree heart block. (Patients with pacemakers may be eligible.)
   * Heart rate <50 bpm during screening.
   * Uncontrolled hypertension (blood pressure >160 mmHg systolic and >100 mmHg diastolic).
2. Patient requires the use of concomitant medications that are contraindicated with cardiac glycosides and/or are known to prolong the QT/QTc interval during study participation (see Appendix 2).
3. Patient has evidence of uncontrolled malabsorptive diarrhea that would prevent adequate absorption of PBI 05204.
4. Patient has dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
5. Patient has uncontrolled or severe intercurrent medical condition (including uncontrolled brain metastases). Patients with stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants are allowed provided there is no dose change within 4 weeks before the first dose of PBI 05204, and no anticipated dose change during study participation.
6. Patient underwent major surgery within 4 weeks before the first dose of PBI 05204 or received cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc.) or an investigational drug or device within 4 weeks (6 weeks for mitomycin C, nitrosoureas, and liposomal doxorubicin) or 5 half-lives of that agent (whichever is shorter) before the first dose of PBI 05204. (For agents in which the total of 5 half-lives is <10 days, there must be a minimum of 10 days between termination of the investigational drug and administration of PBI 05204). Note that prior liver-directed therapies will be permitted (i.e., chemoembolization, radioembolization), as long as target lesions in the liver have demonstrated growth after the liver-directed treatment. Any drug-related toxicity, with the exception of alopecia, should have recovered to ≤ Grade 1.
7. If female, patient is pregnant or breast-feeding.
8. Patient has evidence of a serious active infection (e.g., infection requiring treatment with intravenous antibiotics).
9. Patient has known human immunodeficiency virus (HIV) or hepatitis B or C infection, as such patients may be at increased risk for toxicity due to concomitant treatment, and disease-related symptoms may preclude accurate assessment of the safety of PBI 05204.
10. Patient has an important medical illness or abnormal laboratory finding that, in the Investigator's opinion, would increase the risk of participating in this study.
11. Patient has a history of other malignancy treated with curative intent within the previous 5 years with the exception of adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix. Patients with previous invasive cancers are eligible if the treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
12. Patient was previously exposed to PBI 05204.
13. Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to PBI-05204 (i.e., cardiac glycoside compounds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 4.5 months

SECONDARY OUTCOMES:
Time to Progression | up to 1 year
Time to Treatment Failure | up to 1 year
Progression free survival | up to 1 year
Overall response rate | up to 1 year
Tumor control rate | up to 1 year
Duration of response | up to 1 year
CA 19-9 response | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, MD, Principal Investigator — Vanderbilt University
Locations (5):
- United States (5):
  - Scottsdale Healthcare Hospitals, Scottsdale, Arizona
  - Florida Hospital Tampa, Tampa, Florida
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Roth MT, Cardin DB, Borazanci EH, Steinbach M, Picozzi VJ, Rosemury A, Wadlow RC, Newman RA, Berlin J. A Phase II, Single-Arm, Open-Label, Bayesian Adaptive Efficacy and Safety Study of PBI-05204 in Patients with Stage IV Metastatic Pancreatic Adenocarcinoma. Oncologist. 2020 Oct;25(10):e1446-e1450. doi: 10.1634/theoncologist.2020-0440. Epub 2020 Jul 2. PMID 32452588